CLINICAL TRIAL: NCT04805827
Title: Randomized Single Oral Dose, Open-label, Two-way, Two-periods, Un-replicated Crossover, Bioequivalence Study to Compare Nerpentin600 mg Film Coated Tablet (Gabapentin 600 mg) Manufactured by EGPI (Egyptian Group for Pharmaceutical Industry) - Egypt for Aman Pharma, Versus Neurontin 300 mg Hard Gelatin Capsule (Gabapentin 300 mg) a Product of Pfizer Egypt, Under License From: Parke-Davis-Germany, a Company of Pfizer INC., USA, on Healthy Subjects Under Fasting Condition.
Brief Title: Comparative Randomized, Single Dose, Two-way Crossover Open-label Study to Determine the Bioequivalence of Gabapentin From Nerpentin 600 mg (Test ) F.C.T (Aman Pharma ,Egypt.) and Gabapentin From Neurontin 300 mg (Referance ) H.G.C. ( Pfizer Egypt)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharma Guide CRO (Other)
Responsible Party: Principal Investigator, Mostafa Kaboah, Clinical department manager, Pharma Guide CRO
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PHG-AMA/GAB-0221/01
Record Dates: First submitted 2021-03-13; First posted 2021-03-18 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Pharma Guide; Gabapentin; Neurontin; Mostafa Kaboah
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Randomized single oral dose, open-label, two-way, two-periods, UN-replicated crossover design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): 1 tablet contains 600 mg Gabapentin
  Interventions: Drug: Gabapentin
- Neurontin (Active Comparator): 2 capsule contains 2*300 = 600 mg Gabapentin
  Interventions: Drug: Neurontin

INTERVENTIONS:
Drug: Gabapentin — 1 tablet contains 600 mg Gabapentin
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Neurontin — 2 capsule contains 2*300 = 600 mg Gabapentin
  Arms: Neurontin

SUMMARY:
This study is conducted with the aim to investigate whether any differences concerning the rate and extent of absorption exist between the test and the reference product, Test product was Nerpentine 600 mg Film coated Tablet (Aman Pharma) Reference Product was Neurontin 300 mg Capsule.(Pfizer) The comparative bio availability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

Study was open-label, randomized, crossover, with 02 treatments, 02 sequences and 02 periods, under fasting conditions. one tablet from test product 600 mg against two capsules ( 2*300 mg ) reference product.

Study population was 34 subjects , males ,adults between 18-55 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant female.
2. Subjects should be between the ages of 18 and 55 years.
3. Subject's weight should be within the normal range, preferably have a Body Mass Index between 18.5 and 30 kg/m2.
4. Subjects with normal range of vital signs (Blood Pressure, Pulse Rate.
5. Respiratory Rate and Body Temperature).
6. Normal physical examination at screening visit.
7. Ability to communicate adequately with the investigator himself or his representatives.
8. Ability and agreement to comply with the study requirements.
9. Understanding of the study and agreement to give a written informed consent.
10. The ability of the subjects to understand and comply with the study protocol has to be assessed
11. Females should not be pregnant or lactating.

Exclusion Criteria:

1. Who have a topic constitution or asthma or known allergy for Gabapentin and/or any other ingredients of the products.
2. Symptomatic or asymptomatic orthostatic hypotension at screening or before the first drug administration. Systolic blood pressure less than 100 or more than 140 mm Hg and Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
3. Pulse rate less than 60 pulse/minute or more than 100 pulse/minute.
4. History or presence of significant smoking (≥10 cigarettes or consumption of tobacco products and refusal to restrain from smoking or consumption of tobacco products for 48 hours before dosing until checkout).
5. History of difficulty of donating blood.
6. History of difficulty of swallowing.
7. Any history or presence of clinical relevance of cardiovascular, neurological, musculoskeletal, hematological, hepatic, gastrointestinal, renal, pulmonary, endocraniological, metabolism or psychiatric disease, any type of porphyria.
8. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
9. Participation in a drug research study or donating blood within past 2 months before screening.
10. Subjects who used any of prescribed systemic or topical medication (including OTC medication) within 2 weeks before the initiation of the study (except single doses of analgesics which have no drug interaction with study product).
11. History of allergic response to heparin.
12. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
13. Subjects who regular consumed of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine, chocolate, sodas,) equivalent to more than 500 mg methylxanthines per day, and refusal to abstain from consumption of these products for 48 hours before dosing until checkout).
14. Founding Positive in the alcohol test done at the time of check in.
15. Founding positive in the Urine drugs of abuse at time of check in.
16. Intake of depot injectable solutions (including study medications) within 6 months before start of the study.
17. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before start of the study.
18. Special diet due to any reason, e.g. vegetarian.
19. Subjects who are not suitable to any of inclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of drug gabapentin | 0.0, 0.5, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36 and 48 hours post dose
  (CMAX) Maximum plasma concentration
Area under the plasma concentration versus time curve (AUC) of gabapentin | 0.0, 0.5, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36 and 48 hours post dose
  AUC (Area under the concentration-time curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharma Guide, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 01-04-2021
URL: https://www.pharmaguide-eg.com/